CLINICAL TRIAL: NCT01220492
Title: Phase 1/2 Study of UC-MSC Treatment for the Evaluation the Efficacy and Safety in Patients With Liver Cirrhosis
Brief Title: Umbilical Cord Mesenchymal Stem Cells for Patients With Liver Cirrhosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Fu-Sheng Wang, the Institute of Translational hepatology, Beijing 302 Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: beijing302-002
Record Dates: First submitted 2010-10-04; First posted 2010-10-14 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Liver Cirrhosis
Keywords: liver cirrhosis; mesenchymal stem cells; longer term survival; safety
MeSH Terms: conditions — Liver Cirrhosis | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional plus MSC treatment (Experimental): participants will receive conventional treatment plus a dose of MSC from day 0 through the week 8 study visit. Participants will then be followed until the 75 months study visit.
  Interventions: Drug: conventional plus MSC treatment
- conventional plus placebo treatment (Experimental): participants will receive conventional plus placebo treatment from day 0 through the week 8 study visit. Participants will then be followed until the 75 months study visit.
  Interventions: Drug: conventional plus placebo treatment

INTERVENTIONS:
Drug: conventional plus MSC treatment — received conventional treatment and taken i.v., once per 4 week, at a dose of 0.5*10E6 MSC/kg body for 8 weeks.
  Arms: conventional plus MSC treatment
Drug: conventional plus placebo treatment — received conventional treatment and taken i.v., once per 4 week, at 50 ml saline for 8 weeks.
  Arms: conventional plus placebo treatment

SUMMARY:
Liver cirrhosis (LC) represents a late stage of progressive hepatic fibrosis characterized by distortion of the hepatic architecture and formation of regenerative nodules. The liver transplantation is one of the only effective therapies available to such patients. However, lack of donors, surgical complications, rejection, and high cost are it's serious problems. The potential for stem cells to differentiate into hepatocytes cells was recently confirmed. Particularly, autologous bone marrow-derived mesenchymal stem cell (BM-MSC) has been demonstrated to decrease MELD score and increase serum albumin in the patients with decompensated liver cirrhosis. Therefore, the investigators propose a hypothesis that umbilical cord-derived MSCs (UC-MSC) can also improve the disease conditions of LC patients, particularly reducing the decompensated conditions in these patients.

DETAILED DESCRIPTION:
Liver cirrhosis (LC) represents a late stage of progressive hepatic fibrosis characterized by distortion of the hepatic architecture and formation of regenerative nodules. The liver transplantation is one of the only effective therapies available to such patients. However, lack of donors, surgical complications, rejection, and high cost are it's serious problems.

The potential for stem cells to differentiate into hepatocytes cells was recently confirmed. In particular, bone marrow-derived mesenchymal stem cell (BM-MSC) transplantation has been applicated in the clinic for treat several human diseases such as GVHD, cardiac injury and brain injury, and displayed good tolerance and efficiency. BM-MSC has also been used to treat human liver diseases such as liver failure and liver cirrhosis. In a phase 1 study, autologous BM-MSC transplantation has potential to decrease MELD score and increase serum albumin in the patients with decompensated liver cirrhosis.

The purpose of this study is to learn whether and how umbilical cord-derived MSCs (UC-MSC) can improve the longer term survival in patients with liver cirrhosis. This study will also look at how well BM-MSC is tolerated and its safety in LC patients.

Participants in the study will be randomly assigned to one of two treatment arms:

Arm A: Participants will receive conserved treatment plus three times UC-MSC treatment at 4-week intervals.

Arm B: Participants will receive conserved treatment plus three times saline infusions at 4-week intervals.

UC-MSC will be prepared according to standard procedures and is collected in plastic bags containing anti coagulant. MSCs are infused intravenously. After cell therapy, patients are followed up for 75 months. The evaluation of some clinical parameters such as the level of serum alanine aminotransferase (ALT), total bilirubin (TB),prothrombin time (PT), albumin (ALB), prealbumin(PA), the rountin blood test are detected at week 12, 24, 48 timepoints. Clinical symptoms as well as complication were also observed simultaneously.

ELIGIBILITY:
Inclusion Criteria:

1. Liver cirrhosis
2. Negative pregnancy test (female patients in fertile age)
3. written consent

Exclusion Criteria:

1. Hepatocellular carcinoma or other malignancies
2. Pregnancy
3. sepsis
4. Presence of significant extrahepatic biliary disease (e.g. CBD stone, PSC, etc.)
5. Cardiac, renal or respiratory failure
6. Active thrombosis of the portal or hepatic veins

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
survival time | 75 months
incidence of HCC events | 75 months

SECONDARY OUTCOMES:
The levels of serum albumin | 48 weeks
The levels of serum total bilirubin | 48 weeks
The levels of serum prothrombin activity | 48 weeks
the levels of serum cholinesterase | 48 weeks
complications | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, Professor, Principal Investigator — Beijing 302 Hospital
Locations (1):
- Beijing 302 Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Schuppan D, Afdhal NH. Liver cirrhosis. Lancet. 2008 Mar 8;371(9615):838-51. doi: 10.1016/S0140-6736(08)60383-9. PMID 18328931
- [Background] Kisseleva T, Gigante E, Brenner DA. Recent advances in liver stem cell therapy. Curr Opin Gastroenterol. 2010 Jul;26(4):395-402. doi: 10.1097/MOG.0b013e32833a6bec. PMID 20495456
- [Background] Kharaziha P, Hellstrom PM, Noorinayer B, Farzaneh F, Aghajani K, Jafari F, Telkabadi M, Atashi A, Honardoost M, Zali MR, Soleimani M. Improvement of liver function in liver cirrhosis patients after autologous mesenchymal stem cell injection: a phase I-II clinical trial. Eur J Gastroenterol Hepatol. 2009 Oct;21(10):1199-205. doi: 10.1097/MEG.0b013e32832a1f6c. PMID 19455046
- [Result] Mohamadnejad M, Alimoghaddam K, Mohyeddin-Bonab M, Bagheri M, Bashtar M, Ghanaati H, Baharvand H, Ghavamzadeh A, Malekzadeh R. Phase 1 trial of autologous bone marrow mesenchymal stem cell transplantation in patients with decompensated liver cirrhosis. Arch Iran Med. 2007 Oct;10(4):459-66. PMID 17903050